CLINICAL TRIAL: NCT04052542
Title: Maximizing Extubation Outcomes Through Educational and Organizational Research: Think NIV Pilot Study
Brief Title: METEOR Think NIV Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Timothy Girard, MD, MSCI, Associate Professor, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY19050064; U01HL143507 (NIH)
Record Dates: First submitted 2019-08-08; First posted 2019-08-09 (Actual); Results first posted 2021-09-17 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Acute Respiratory Failure
Keywords: Noninvasive ventilation; Education; Intensive care unit; Mechanical ventilation; Evidence-based practice

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional online continuing education (Active Comparator)
  Interventions: Behavioral: Traditional online continuing education
- Interprofessional education (Active Comparator)
  Interventions: Behavioral: Interprofessional education
- Just-in-time education (Active Comparator)
  Interventions: Behavioral: Just-in-time education

INTERVENTIONS:
Behavioral: Traditional online continuing education — 30-minute, online, interactive, educational video describing the benefits of preventive post-extubation NIV, the indications and contraindications for preventive post-extubation NIV, and the value of working together as an interprofessional ICU team when implementing preventive post-extubation NIV
  Arms: Traditional online continuing education
Behavioral: Interprofessional education — One-time, 90-120-minute, in-person, interprofessional educational workshop consisting of a 30-minute didactic session and a 60-90-minute small group session
  Arms: Interprofessional education
Behavioral: Just-in-time education — "Just-in-time," point-of-care education provided by trained advanced practice providers who will be on-hand in the study ICU, where they will deliver the education at the bedside during rounds when a patient meets criteria for preventive post-extubation NIV
  Arms: Just-in-time education

SUMMARY:
This study will pilot test three strategies designed to speed implementation of preventive post-extubation noninvasive ventilation (NIV): one control strategy (traditional online continuing medical education) and two novel strategies (interprofessional education and just-in-time education).

DETAILED DESCRIPTION:
During a one-month intervention period, the investigators will pilot test the educational strategies in three participating UPMC ICUs. Prior to receiving education, participants will be invited to complete a short online survey. Participants in the control group will be invited to complete a 30-minute online continuing education module, which will conclude with a survey. Participants in the interprofessional education group will be invited to attend a 90-minute, in-person, interprofessional education session that will occur in or near the participating ICU. A trained advance practice provider will provide participants in the just-in-time education group with 5-10 minutes of education in the ICU when the ICU team is rounding on a patient who is identified to be high risk for extubation failure. The just-in-time education may occur more than once per day, depending on the number of high-risk patients identified. All educational strategies will include content on the benefits of preventive post-extubation NIV, the indications and contraindications for preventive post-extubation NIV, and the value of working together as an interprofessional ICU team when implementing preventive post-extubation NIV. Each educational intervention will include a survey designed to determine the feasibility, acceptability, and preliminary impact of the educational strategies. The investigators will also directly observe instances of interprofessional and just-in-time education and conduct in-person interviews to assess these factors in a qualitative manner. Lastly, during the intervention period and the 6 months before and after the intervention period, the investigators will collect data from the electronic health record and analyze changes in percent of high-risk patients who receive preventive post-extubation NIV, reintubation rate, duration of mechanical ventilation, ventilator-associated pneumonia, and in-hospital mortality.

ELIGIBILITY:
Two study populations will be included.

Learners (population 1) will include:

* frontline care providers, including physicians, advanced practice providers, nurses, and respiratory therapists
* working in a participating ICU.

Frontline care providers will be excluded if they:

* have not worked in their current UPMC ICU for more than one month prior to the current study
* have not directly cared for a mechanically ventilated patient in a UPMC ICU during the three months preceding the current study.

Patients (population 2) will include:

* mechanically ventilated patients
* treated in the participating ICUs
* surviving to extubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1328 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy D Girard, MD, MSCI, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Thille AW, Harrois A, Schortgen F, Brun-Buisson C, Brochard L. Outcomes of extubation failure in medical intensive care unit patients. Crit Care Med. 2011 Dec;39(12):2612-8. doi: 10.1097/CCM.0b013e3182282a5a. PMID 21765357
- [Background] Ferrer M, Sellares J, Valencia M, Carrillo A, Gonzalez G, Badia JR, Nicolas JM, Torres A. Non-invasive ventilation after extubation in hypercapnic patients with chronic respiratory disorders: randomised controlled trial. Lancet. 2009 Sep 26;374(9695):1082-8. doi: 10.1016/S0140-6736(09)61038-2. Epub 2009 Aug 12. PMID 19682735
- [Background] Ouellette DR, Patel S, Girard TD, Morris PE, Schmidt GA, Truwit JD, Alhazzani W, Burns SM, Epstein SK, Esteban A, Fan E, Ferrer M, Fraser GL, Gong MN, Hough CL, Mehta S, Nanchal R, Pawlik AJ, Schweickert WD, Sessler CN, Strom T, Kress JP. Liberation From Mechanical Ventilation in Critically Ill Adults: An Official American College of Chest Physicians/American Thoracic Society Clinical Practice Guideline: Inspiratory Pressure Augmentation During Spontaneous Breathing Trials, Protocols Minimizing Sedation, and Noninvasive Ventilation Immediately After Extubation. Chest. 2017 Jan;151(1):166-180. doi: 10.1016/j.chest.2016.10.036. Epub 2016 Nov 3. PMID 27818331
- [Background] Rochwerg B, Brochard L, Elliott MW, Hess D, Hill NS, Nava S, Navalesi P Members Of The Steering Committee, Antonelli M, Brozek J, Conti G, Ferrer M, Guntupalli K, Jaber S, Keenan S, Mancebo J, Mehta S, Raoof S Members Of The Task Force. Official ERS/ATS clinical practice guidelines: noninvasive ventilation for acute respiratory failure. Eur Respir J. 2017 Aug 31;50(2):1602426. doi: 10.1183/13993003.02426-2016. Print 2017 Aug. PMID 28860265

RESULTS

PARTICIPANT FLOW:
Groups:
- Traditional Online Continuing Education Group - Pre-education: Patients admitted during the 6 months prior to the education period to the ICU that would later participate in traditional online continuing education.
- Traditional Online Continuing Education Group - During Education: Patients admitted during the one-month education period to the ICU that participated in traditional online continuing education.
- Traditional Online Continuing Education Group - Post-education: Patients admitted during the 6 months after the education period to the ICU that participated in traditional online continuing education.
- Interprofessional Education Group - Pre-education: Patients admitted during the 6 months prior to the education period to the ICU that would later participate in interprofessional education.
- Interprofessional Education - During Education: Patients admitted during the one-month education period to the ICU that participated in interprofessional education.
- Interprofessional Education Group - Post-education: Patients admitted during the 6 months after the education period to the ICU that participated in interprofessional education.
- Just-in-time Education - Pre-education: Patients admitted during the 6 months prior to the education period to the ICU that would later participate in just-in-time education.
- Just-in-time Education Group - During Education: Patients admitted during the one-month education period to the ICU that participated in just-in-time education.
- Just-in-time Education Group - Post-education: Patients admitted during the 6 months after the education period to the ICU that participated in just-in-time education.
- Traditional Online Continuing Education Group - Learners: Learners who participated in traditional online continuing education
- Interprofessional Education Group - Learners: Learners who participated in interprofessional education
- Just-in-time Education Group - Learners: Learners who participated in just-in-time education
Period: Overall Study
Arm/Group | Traditional Online Continuing Education Group - Pre-education | Traditional Online Continuing Education Group - During Education | Traditional Online Continuing Education Group - Post-education | Interprofessional Education Group - Pre-education | Interprofessional Education - During Education | Interprofessional Education Group - Post-education | Just-in-time Education - Pre-education | Just-in-time Education Group - During Education | Just-in-time Education Group - Post-education | Traditional Online Continuing Education Group - Learners | Interprofessional Education Group - Learners | Just-in-time Education Group - Learners
Started | 116 | 28 | 146 | 188 | 24 | 183 | 275 | 27 | 276 | 22 | 31 | 12
Completed | 116 | 28 | 146 | 188 | 24 | 183 | 275 | 27 | 276 | 22 | 31 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Traditional Online Continuing Education Group - Pre-education | Traditional Online Continuing Education Group - During Education | Traditional Online Continuing Education Group - Post-education | Interprofessional Education Group - Pre-education | Interprofessional Education - During Education | Interprofessional Education Group - Post-education | Just-in-time Education - Pre-education | Just-in-time Education Group - During Education | Just-in-time Education Group - Post-education | Traditional Online Continuing Education Group - Learners | Interprofessional Education Group - Learners | Just-in-time Education Group - Learners | Total
Number analyzed (Participants) | 116 | 28 | 146 | 188 | 24 | 183 | 275 | 27 | 276 | 22 | 31 | 12 | 1328
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Baseline characteristics were collected and analyzed only for patient participants. The characteristics of learner participants were not recorded.
  years
    number analyzed (Participants) | 116 | 28 | 146 | 188 | 24 | 183 | 275 | 27 | 276 | 0 | 0 | 0 | 1263
    (all) | 72 [68 to 77] | 79 [72 to 84] | 74 [70 to 80] | 74 [70 to 79] | 77 [72 to 79] | 75 [70 to 78] | 70 [69 to 77] | 69 [68 to 71] | 71 [69 to 77] |  |  |  | 73 [69 to 77]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline characteristics were collected and analyzed only for patient participants. The characteristics of learner participants were not recorded.
  Participants
    number analyzed (Participants) | 116 | 28 | 146 | 188 | 24 | 183 | 275 | 27 | 276 | 0 | 0 | 0 | 1263
    Female | 52 | 20 | 71 | 85 | 10 | 100 | 165 | 7 | 87 |  |  |  | 597
    Male | 64 | 8 | 75 | 103 | 14 | 83 | 110 | 20 | 189 |  |  |  | 666
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Baseline characteristics were collected and analyzed only for patient participants. The characteristics of learner participants were not recorded.
  Participants
    Race: number analyzed (Participants) | 116 | 28 | 146 | 188 | 24 | 183 | 275 | 27 | 276 | 0 | 0 | 0 | 1263
    Race: White | 96 | 23 | 120 | 177 | 23 | 170 | 236 | 21 | 186 |  |  |  | 1052
    Race: Black | 10 | 2 | 20 | 6 | 0 | 7 | 20 | 4 | 56 |  |  |  | 125
    Race: Other | 10 | 3 | 6 | 5 | 1 | 6 | 19 | 2 | 34 |  |  |  | 86
Sequential Organ Failure Assessment (SOFA) Score [Median (Inter-Quartile Range); unit: units on a scale] — The Sequential Organ Failure Assessment (SOFA) score is a validated tool that quantifies the number and severity of failed organs. Higher scores indicate worse organ failure. Minimum = 0; maximum = 24. Population: The Sequential Organ Failure Assessment (SOFA) score does not apply to learner participants.
  units on a scale
    number analyzed (Participants) | 116 | 28 | 146 | 188 | 24 | 183 | 275 | 27 | 276 | 0 | 0 | 0 | 1263
    (all) | 9 [6 to 11] | 7 [6 to 9] | 7 [4 to 9] | 8 [5 to 10] | 9 [8 to 10] | 8 [6 to 11] | 7 [4 to 9] | 10 [5 to 13] | 5 [4 to 8] |  |  |  | 7 [4 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Number of ICU Team Members (Learners) Who Received Education
Description: This implementation outcome measuring reach only applies to learner participants.
Time Frame: Up to 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Traditional Online Continuing Education Group - Learners | Interprofessional Education Group - Learners | Just-in-time Education Group - Learners
Number analyzed (Participants) | 22 | 31 | 12
Participants | 22 | 31 | 12

2. Primary Outcome: Learner Attitudes Regarding Education (Mean Scores on Relevant Survey Questions)
Description: Using a 5-point Likert scale (1=strongly disagree; 5=strongly agree), learners reported their level of agreement with the statement "I liked the way the information was presented." This outcome only applies to learner participants.
Time Frame: Up to 10 weeks
Population: The Overall Number of Participants Analyzed is not consistent with numbers provided in the Participant Flow module because some learner participants did not complete the survey the assessed this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Traditional Online Continuing Education Group - Learners | Interprofessional Education Group - Learners | Just-in-time Education Group - Learners
Number analyzed (Participants) | 14 | 30 | 12
score on a scale | 4.2 (0.7) | 4.8 (0.6) | 3.4 (1.0)

3. Secondary Outcome: Number of High-risk Patients Without Contraindications Who Received Post-extubation Noninvasive Ventilation
Description: This implementation outcome only applies to patient participants.
Time Frame: Participants will be followed for the duration of their hospital admission, estimated to be 1-2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Traditional Online Continuing Education Group - Pre-education | Traditional Online Continuing Education Group - During Education | Traditional Online Continuing Education Group - Post-education | Interprofessional Education Group - Pre-education | Interprofessional Education - During Education | Interprofessional Education Group - Post-education | Just-in-time Education - Pre-education | Just-in-time Education Group - During Education | Just-in-time Education Group - Post-education
Number analyzed (Participants) | 116 | 28 | 146 | 188 | 24 | 183 | 275 | 27 | 276
Participants | 2 | 2 | 2 | 0 | 1 | 1 | 4 | 1 | 5

4. Secondary Outcome: Learner Role Clarity (Mean Scores on Relevant Survey Questions)
Description: Using a 5-point Likert scale (1=strongly disagree; 5=strongly agree), learners reported their level of agreement with the statement "In assessing mechanically ventilated patients for potential extubation, I know what my responsibilities are." This outcome only applies to learner participants.
Time Frame: Up to 10 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Traditional Online Continuing Education Group - Learners | Interprofessional Education Group - Learners | Just-in-time Education Group - Learners
Number analyzed (Participants) | 14 | 30 | 12
score on a scale | 4.2 (0.7) | 4.9 (0.3) | 4.8 (0.4)

5. Secondary Outcome: Learner Specialization (Mean Scores on Relevant Survey Questions)
Description: Using a 5-point Likert scale (1=strongly disagree; 5=strongly agree), learners reported their level of agreement with the statement "In assessing mechanically ventilated patients for potential extubation, I have knowledge that no other team member has." This outcome only applies to learner participants.
Time Frame: Up to 10 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Traditional Online Continuing Education Group - Learners | Interprofessional Education Group - Learners | Just-in-time Education Group - Learners
Number analyzed (Participants) | 14 | 30 | 12
score on a scale | 3.6 (1.1) | 3.4 (1.3) | 3.3 (1.2)

6. Secondary Outcome: Learner Credibility (Mean Scores on Relevant Survey Questions)
Description: Using a 5-point Likert scale (1=strongly disagree; 5=strongly agree), learners reported their level of agreement with the statement "In making decisions about extubation, I am comfortable accepting procedural suggestions from other team members." This outcome only applies to learner participants.
Time Frame: Up to 10 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Traditional Online Continuing Education Group - Learners | Interprofessional Education Group - Learners | Just-in-time Education Group - Learners
Number analyzed (Participants) | 14 | 30 | 12
score on a scale | 4.5 (0.7) | 4.9 (0.3) | 4.7 (0.5)

7. Secondary Outcome: Learner Coordination (Mean Scores on Relevant Survey Questions)
Description: Using a 5-point Likert scale (1=strongly disagree; 5=strongly agree), learners reported their level of agreement with the statement "In delivering care to patients in respiratory failure, our ICU team works together in a well-coordinated fashion." This outcome only applies to learner participants.
Time Frame: Up to 10 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Traditional Online Continuing Education Group - Learners | Interprofessional Education Group - Learners | Just-in-time Education Group - Learners
Number analyzed (Participants) | 14 | 30 | 12
score on a scale | 4.3 (0.7) | 4.9 (0.3) | 4.3 (0.9)

8. Secondary Outcome: Learner Psychological Safety (Mean Scores on Relevant Survey Questions)
Description: Using a 5-point Likert scale (1=strongly disagree; 5=strongly agree), learners reported their level of agreement with the statement "I'm confident that when I make suggestions, other members of the care team will listen." This outcome only applies to learner participants.
Time Frame: Up to 10 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Traditional Online Continuing Education Group - Learners | Interprofessional Education Group - Learners | Just-in-time Education Group - Learners
Number analyzed (Participants) | 14 | 30 | 12
score on a scale | 3.9 (0.7) | 4.6 (0.5) | 4.7 (0.5)

9. Secondary Outcome: Learner Perspectives on Leader Inclusiveness (Mean Scores on Relevant Survey Questions)
Description: Using a 5-point Likert scale (1=strongly disagree; 5=strongly agree), learners reported their level of agreement with the statement "From now on, physicians in this ICU are likely to strike an appropriate balance between authority and openness to suggestion." This outcome only applies to learner participants.
Time Frame: Up to 10 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Traditional Online Continuing Education Group - Learners | Interprofessional Education Group - Learners | Just-in-time Education Group - Learners
Number analyzed (Participants) | 14 | 30 | 12
score on a scale | 3.9 (0.5) | 4.7 (0.5) | 4.2 (0.9)

ADVERSE EVENTS:
Time Frame: In-hospital, up to 60 days
Description: In-hospital adverse events only apply to patient groups. All-cause mortality, serious adverse events, and other (not including serious) adverse events were not monitored in the learner groups because participation involved minimal risk for learners.
Arm/Group | Traditional Online Continuing Education Group - Pre-education | Traditional Online Continuing Education Group - During Education | Traditional Online Continuing Education Group - Post-education | Interprofessional Education Group - Pre-education | Interprofessional Education - During Education | Interprofessional Education Group - Post-education | Just-in-time Education - Pre-education | Just-in-time Education Group - During Education | Just-in-time Education Group - Post-education | Traditional Online Continuing Education Group - Learners | Interprofessional Education Group - Learners | Just-in-time Education Group - Learners
All-Cause Mortality (participants affected / at risk) | 44/116 | 10/28 | 61/146 | 37/188 | 8/24 | 58/183 | 130/275 | 5/27 | 57/276 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/116 | 0/28 | 0/146 | 0/188 | 0/24 | 0/183 | 0/275 | 0/27 | 0/276 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/116 | 0/28 | 0/146 | 0/188 | 0/24 | 0/183 | 0/275 | 0/27 | 0/276 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
By design, this was a non-randomized pilot trial intended to assess the feasibility, acceptability, and preliminary impact of three strategies designed to speed implementation of post-extubation noninvasive ventilation among high-risk patients recovering from acute respiratory failure. The effects of the educational interventions on patient outcomes cannot be reliably determined using data from this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT04052542/Prot_SAP_000.pdf